CLINICAL TRIAL: NCT02278172
Title: The Effects of Vitamin D Supplementation on VO2max in Athletes: a Randomised, Double-blind, Placebo-controlled Trial
Brief Title: The Effects of Vitamin D Supplementation on Aerobic Fitness in Athletes
Acronym: VDAF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Ulster (Other)
Collaborators: Northern Ireland Executive (Unknown)
Responsible Party: Principal Investigator, Dr Pamela Magee, Dr Pamela Magee, University of Ulster
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: REC14.0087
Record Dates: First submitted 2014-10-27; First posted 2014-10-29 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Aerobic Fitness (VO2max)
Keywords: vitamin D; athletes; fitness
MeSH Terms: interventions — Vitamin D; Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Vitamin D3 3000IU (75μg) (Active Comparator): Treatment solution delivered via oral spray once daily for 12-weeks
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator): Placebo solution delivered via oral spray once daily for 12-weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D — 3000IU (75 μg) vitamin D in a commercially available oral spray solution
  Other Names: cholecalciferol; vitamin D3
  Arms: Vitamin D3 3000IU (75μg)
Dietary Supplement: Placebo — Placebo oral spray solution manufactured to mimic the vitamin D oral spray
  Arms: Placebo

SUMMARY:
The primary aim of the study is to identify if vitamin D3 supplementation influences VO2max in athletes.

Secondary aims are to determine if vitamin D3 supplementation impacts on measures of muscle function, lung function, body composition, immune function and the self-reported incidence of upper respiratory tract infection.

This double-blind, randomised, placebo-controlled trial is of parallel design and will aim to recruit a total of 50 athletes randomised into either a placebo or treatment group for a 12-week intervention.

ELIGIBILITY:
Inclusion Criteria:

* Athletes whose sport does not primarily consist of an anaerobic component
* Apparently healthy
* Over the age of 18

Exclusion Criteria:

* Resting arterial hypertension
* Individuals who are not an athlete at a University/local sports team
* Athletes who predominantly utilise anaerobic energy systems
* Athletes under the age of 18
* Those that have consumed a supplement containing vitamin D (greater than 400IU/day) or iron supplements for up to 30 days prior to starting the study
* Those with health conditions identified by the screening questionnaire
* Individuals that are on prescribed medication that is known to affect vitamin D metabolism
* Those following a vegan diet
* Those with a physical disability that would prevent successful completion of the exercise test
* Those who have either had a sun holiday in the 4 weeks prior to starting the study
* Those planning a sun holiday during the intervention period

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Aerobic fitness (VO2max) | At baseline and at 12-weeks
  A medical screening questionnaire will be completed prior to the test. Athletes resting blood pressure will be measured twice to rule out resting hypertension. After a standardised warm-up, starting speed will be 8/km/hr at 1% incline, until 17/km/hr, after which incline will increase by 1% every minute until VO2max is met. A metabolic cart (Metalyzer 3B) will measure the athlete's ventilation (oxygen uptake and carbon dioxide output) throughout the test.
  The test will be terminated when two of the following criterion are met*:
  Respiratory exchange ratio reaches/exceeds 1.15 AND VO2 plateau observed OR Heart rate within 10bpm of age-predicted maximum
  * Except when volitional exhaustion occurs Athletes will be asked to refrain from strenuous activity for 24 hours prior to VO2max testing in order to control for last bout effects.
  Post-exercise lactate concentration (age and gender adjusted) will further-verify that VO2max was attained using a Lactate Pro device.

SECONDARY OUTCOMES:
Hand grip strength | At baseline and at 12-weeks
  Hand grip dynamometry will be used to assess athletes grip strength. This will be measured on both dominant and non-dominant hands three times. The athlete will be asked to hold the device and grip as tightly as possible whilst holding the device alongside their body. There will be a 10 second rest period between measurements.
Vertical jump height | At baseline and at 12-weeks
  Athletes will be asked to reach upwards as far as possible, from a standing position and mark this point on a wall. After this they will be asked to perform a counter-movement jump a total of 3 times with a 10 second rest-period between jumps, reaching as high as possible and making a mark each time. Vertical jump height is calculated from the difference between standing reach height and the best height reached when performing a counter-movement jump.
Lung function | At baseline and at 12-weeks
  Forced expiratory volume at 1 second (FEV1) and forced vital capacity (FVC) will be measured. A calibrated Carefusion® MicroLab portable spirometer will be used to measure these variables.The athletes will need to take a maximal inhalation and then perform a full exhalation as fast as possible into a disposable mouthpiece.
  This procedure will be repeated three times and an average taken at each time-point. The timing of repeats will be at the athletes discretion.
Nutrient intake | At baseline only/ at baseline and at 12-weeks
  Dietary vitamin D and calcium intake will be estimated using a validated food frequency questionnaire at one time point (baseline only). This is due to studies highlighting equivocal variation in dietary vitamin D intake throughout the year.
  24hr recalls will be completed at baseline and at 12-weeks in order to derive mean nutrient intakes for the vitamin D and placebo treatment groups respectively.
Self-reported upper respiratory illness | Once per week up to week 12
  An online questionnaire will allow athletes to record if they have any symptoms that are associated with upper respiratory infections. The athlete will be asked to mark a series of boxes to indicate how many symptom(s) if any that they have had each week.
Physical activity levels | At baseline and at 12-weeks
  The 'Modified Recent Physical Activity Questionnaire' produced by the Medical Research Council (a validated physical activity questionnaire) will be completed on two occasions to estimate physical activity levels.
Body composition | At baseline and at 12-weeks
  Body composition will be measured using the BodPod, employing air plethysmography (displacement of air) to accurately measure percentage fat mass and percentage fat-free mass.
Vitamin D status | At baseline and at 12-weeks
  25-hydroxyvitamin D (25(OH)D) will be quantified, in serum, using liquid chromatography-tandem mass spectrometry (LCMS/MS). Other biomarkers of vitamin D metabolism (adjusted calcium and parathyroid hormone) will be quantified using a clinical chemistry analyser and commercially available enzyme-linked immunosorbent assay.
Immune function | At baseline and at 12-weeks
  A range of immune markers such as interleukin-6, cathelicidin (LL-37) and C-reactive protein will be measured using a commercially available multiplex immunoassay.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela J Magee, PhD, Principal Investigator — University of Ulster
Locations (1):
- Human Intervention Studies Unit (HISU), University of Ulster, Coleraine, Londonderry, United Kingdom